CLINICAL TRIAL: NCT03046641
Title: The Study of Various Models of Exercise Duration on Weight Loss and Lipid Profile in Sedentary Overweight/Obese Middle-aged Men
Brief Title: Exercise Duration Models, in Middle-aged Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P.L.Shupik National Medical Academy of Post-Graduate Education (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, MD, PhD, sports medicine (sports injury and corrective movement), University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No Grant-2
Record Dates: First submitted 2013-06-21; First posted 2017-02-08 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Weight Loss
Keywords: Caloric Restriction; Dietary Formulations; Exercise; Men
MeSH Terms: conditions — Weight Loss; Motor Activity; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous training group (Experimental): With the continuous training program
  Interventions: Other: Continuous training
- interval training group (Experimental): With the interval training program
  Interventions: Other: The interval training

INTERVENTIONS:
Other: Continuous training — Study group I (42 participants) received the continuous training.
  Other Names: group I
  Arms: continuous training group
Other: The interval training — Study group II (40 participants) received the interval training.
  Other Names: group II
  Arms: interval training group

SUMMARY:
Duration of exercise is an important factor among the medical guides for weight loss. However, there is still little knowledge about other its models in middle-aged and older men. The present study aimed to determine the effects of the interval training on weight loss and lipid profile, and to compare its efficiency with the continuous training.

DETAILED DESCRIPTION:
Participants included sedentary men (age 45-75 years) with overweight or obesity (n= 82). They were randomly divided into two groups including continuous exercise, and interval exercise. The weight assessment parameters including change in weight and body composition, blood sample tests were performed pre- and three month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle
* Good Health
* Weight stability

Exclusion Criteria:

Abnormality or history of Disease

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
4-item | 3 months
  weight, lipid profile (HDL, LDL, Cholesterol)

SECONDARY OUTCOMES:
4-item | 3 months
  weight, lipid profile (HDL, LDL, Cholesterol)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Rezaeipour, M.D., PhD., Principal Investigator — Member of Scientific Board in Physical Education and Sport Sciences of Sistan and Baluchestan University

IPD SHARING:
Plan to Share IPD: No